CLINICAL TRIAL: NCT01866488
Title: The Obstetric Cook Double Balloon Catheter in Combination With Oral Misoprostol for Induction of Labor: A Double-Blinded, Randomized Controlled Trial
Brief Title: The Obstetric Cook Double Balloon Catheter in Combination With Oral Misoprostol for Induction of Labor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Meg Hill, Fellow, Maternal Fetal Medicine, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-1027-01
Record Dates: First submitted 2013-04-30; First posted 2013-05-31 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Labor Induction
Keywords: Labor induction; Misoprostol; Cytotec; Cook Obstetric Double Balloon Catheter
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cook Catheter, Oral Misoprostol (Experimental): Cook Catheter is placed and a 50mcg misoprostol tablet is given orally. A repeat dose is administered in 3 hours.
  Interventions: Drug: Misoprostol
- Cook Catheter, Oral Placebo (Placebo Comparator): Cook Catheter is placed and a placebo tablet is given orally. A repeat dose is administered in 3 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Cytotec
  Arms: Cook Catheter, Oral Misoprostol
Other: Placebo
  Arms: Cook Catheter, Oral Placebo

SUMMARY:
The current study is a randomized, controlled, double-blinded trial of Obstetric Cook Catheter combined with oral misoprostol for induction of labor in pregnant patients. The primary outcome to be studied is vaginal delivery rate for the Obstetric Cook Catheter in combination with oral placebo and the Obstetric Cook Catheter in combination with oral misoprostol. Secondary outcomes to be studied include the safety of the method, composite maternal morbidity and composite neonatal morbidity.

The hypothesis is that there is a higher vaginal delivery rate in the patient whom receive both the Obstetric Cook Catheter and the oral misoprostol.

ELIGIBILITY:
Inclusion Criteria:

1. Single, live fetus
2. Cephalic (head-first) presentation
3. Reassuring fetal health assessment
4. Gestational age between 23 and 42 weeks
5. Maternal age 18 and above
6. Bishop score less than 8 in primigravidae
7. Bishop score less than 6 in multigravidae

Exclusion Criteria:

1. Fetal demise 2. Fetal malpresentation 3. Estimated fetal weight less than 500 grams or more than 4000 grams 4. Placenta previa 5. Non-reassuring fetal health assessment 6. Active maternal asthma exacerbation requiring additional medications from the usual medication requirements.

7. History of cesarean section 8. Rupture of amniotic membrane 9. Latex allergy 10. Spontaneous labor 11. Other contraindication to vaginal delivery 12. Allergy to misoprostol of cook catheter

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Occurence of cesarean section | Within 96 hours from the commencement of the Induction of Labor

SECONDARY OUTCOMES:
Time from start of induction of labor to vaginal delivery | 24, 48 and 72 hours

OTHER OUTCOMES:
Change in cervical bishop score with allotted treatment | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Meg Hill, MBBS, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264